CLINICAL TRIAL: NCT06057467
Title: Early Versus Late Initiation of Anticoagulation in Mild-to-moderate Acute Ischemic Stroke Patients With Non-valvular Atrial Fibrillation
Brief Title: Early Versus Late Initiation of Anticoagulation in Mild-to-moderate AIS Patients With NVAF
Acronym: ASAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ASAP
Record Dates: First submitted 2023-09-13; First posted 2023-09-28 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-09

CONDITIONS: Acute Ischemic Stroke; Atrial Fibrillation
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation | interventions — Anticoagulants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early initiation of anticoagulation (Experimental): For patients with NIHSS 0-3, anticoagulation therapy will be initiated within 0-3 days of onset.
  For patients with NIHSS 4-8, anticoagulation therapy will be initiated within 4-6 days of onset.
  Interventions: Drug: Anticoagulation Agents
- Late initiation of anticoagulation (Active Comparator): For patients with NIHSS 0-3, anticoagulation therapy will be initiated within 4-12 days of onset.
  For patients with NIHSS 4-8, anticoagulation therapy will be initiated within 7-12 days of onset.
  Interventions: Drug: Anticoagulation Agents

INTERVENTIONS:
Drug: Anticoagulation Agents — Anticoagulation agents includes rivaroxaban, dabigatran, apixaban, and edoxaban.

SUMMARY:
The goal of this clinical trial is to compare the effectiveness between early and late initiation of anticoagulation therapy in acute ischemic stroke (AIS) patients with non-valvular atrial fibrillation (NVAF). Participants will be 1:1 randomized into early or late initiation group. The primary endpoint is early neurological deterioration (END) before discharge.

DETAILED DESCRIPTION:
Anticoagulation therapy is effective to prevent ischemic stroke in patients with NVAF who have a history of stroke. Recent clinical trials have demonstrated that early initiation of anticoagulation therapy after AIS is safe, while no remarkable benefits have been observed. The goal of this clinical trial is to compare the effectiveness between early and late initiation of anticoagulation therapy in AIS patients with non-NVAF. Participants will be 1:1 randomized into early or late initiation group. The primary endpoint is END before discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Acute ischemic stroke with onset < 48 hours
* Have a history or newly diagnosed as NVAF
* NIHSS on admission <= 8

Exclusion Criteria:

* Chronic renal dysfunction (GFR < 30ml/min) or severe hepatic injury
* Have a history or newly diagnosed as valvular heart disease
* Mural thrombus in heart
* Contraindications of anticoagulation therapy within 12 days after AIS, e.g. severe intracranial hemorrhage
* Received reperfusion therapy, e.g. intravenous thrombolysis and endovascular treatment
* Concomitant stenosis (>50%) of carotid artery/intracranial artery, of which the ischemic lesion located within the territory
* Life expectancy less than 1 year
* Plan to receive invasive surgery in the following 3 months and have high risk of uncontrollable bleeding
* Pregnant or lactating women
* Individuals identified by researchers as unsuitable for participation in the study due to other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2351 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Early neurological deterioration before discharge | At discharge, an average of 7 days
  NIHSS at discharge increase at least 2 points compared with NIHSS on admission

SECONDARY OUTCOMES:
90-day Composite events | 90 days
  Composite events including ischemic stroke, hemorrhagic stroke, myocardial infarction, systemic embolism, major extracranial hemorrhage, and vascular death within 90 days after enrollment
90-day ischemic stroke | 90 days
  Ischemic stroke within 90 days after enrollment
90-day hemorrhagic stroke | 90 days
  Hemorrhagic stroke within 90 days after enrollment
90-day myocardial infarction | 90 days
  Myocardial infarction within 90 days after enrollment
90-day systemic embolism | 90 days
  Systemic embolism within 90 days after enrollment
90-day major extracranial hemorrhage | 90 days
  Major extracranial hemorrhage within 90 days after enrollment
90-day non-major bleeding | 90 days
  Non-major bleeding within 90 days after enrollment
90-day vascular death | 90 days
  Vascular death within 90 days after enrollment
90-day all-cause death | 90 days
  All-cause death within 90 days after enrollment
Discharge mRS | At discharge, an average of 7 days
  Modified Rankin scale at discharge

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou
  - Jiaxing Second Hospital, Jiaxing

IPD SHARING:
Plan to Share IPD: No